CLINICAL TRIAL: NCT03931239
Title: An Open Label, Multicentric, Bridging Study to Assess the Safety of Diphtheria, Tetanus, Pertussis, Hepatitis B and Haemophilus Influenzae Type b Conjugate Vaccine (Adsorbed) Manufactured by Serum Institute of India Pvt. Ltd in Vietnamese Infants Aged 6-12 Weeks, Given as a 3-dose Regime, With 4 Week Intervals Between the Doses
Brief Title: The Transparent Safety Study of the 5 in 1 (DTwP-rHepB-Hib) Combination Vaccine Produced by the Indian Serine Institute in Children of Viet Nam Healthy From 6 to 12 Weeks of Age in a 3-dose Regimen, the Interval Between Doses is 4 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vabiotech (Industry)
Collaborators: Vietstar Biomedical Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VABIOTECH-01
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus Influenzae Type B
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Haemophilus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccination (Experimental): DTPw-HB-Hib vaccine
  Interventions: Biological: Study subjects will be vaccinated with 3 (three) vaccine doses. The first vaccine will be administered intramuscularly starting at 6-12 weeks of age followed by two doses at four-week interval

INTERVENTIONS:
Biological: Study subjects will be vaccinated with 3 (three) vaccine doses. The first vaccine will be administered intramuscularly starting at 6-12 weeks of age followed by two doses at four-week interval — An openlabel, multicentric, bridging study to assess the safety of Diphtheria, Tetanus, Pertussis, Hepatitis B and Haemophilus influenzae type b Conjugate Vaccine (Adsorbed) manufactured by Serum Institute of India Pvt. Ltd in Vietnamese infants aged 6-12 weeks, given as a 3-dose regime, with 4 week intervals between the doses

SUMMARY:
The objective of this study is to evaluate safety and tolerability of Diphtheria, Tetanus, Pertussis, Hepatitis B and Haemophilus influenzae type b Conjugate Vaccine Adsorbed in Vietnamese infants aged 6-12 weeks. This is an open label, single group, bridging study.

DETAILED DESCRIPTION:
This will be an open label, single group, bridging study. Study subjects will be vaccinated with 3 (three) vaccine doses. The first vaccine will be administered intramuscularly starting at 6-12 weeks of age followed by two doses at four-week interval.

This study was performed in strict accordance with Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants, both sexes, between 6 and 12 weeks of age on the day of screening and enrollment
* Subject born at full term of pregnancy (greater or equal to 37 weeks) and Birth weight ≥2500 grams
* Weight ≥ 3,300 grams at the time of screeningSubject with good health as determined by the medical history, physical examination and clinical judgment of the Investigator
* Parent / legal representative can understand and be able to comply with the requirements of the protocol
* Subjects born to mothers who are seronegative to HIV, HBV and HCV through a blood test or maternity record.
* Parent / legal representative is willing to voluntarily sign the consent form for the participant

Exclusion Criteria:

* History of diphtheria, tetanus, pertussis, hepatitis B, or Hib infections (confirmed either clinically, serologically or microbiologically)
* Fever (temperature ≥37.50C) or hypothermia (≤35.50C) or acute illness / infection that requires treatment.
* Previous vaccination against diphtheria, tetanus, pertussis and Haemophilus influenzae type b diseases.
* Known allergy to any component of the vaccine;
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination.
* Being treated with anticoagulants or at high risk of bleeding.
* A family history of SIDS (sudden infant death syndrome)
* Have received any blood products, corticosteroids, cytotoxic drugs, immunosuppressive therapy, radiation therapy in the last 4 weeks.
* Have participated in another clinical trial within 30 days prior to the study vaccination or may participate in the course of the study.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects.
* History of any neurological disorders or seizures

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Percent of Participants With Adverse Events Related to DTPw-HB-Hib vaccine Administration | Days 0 to 28 post-vaccination

SECONDARY OUTCOMES:
Percent of Participants With Adverse Events Related to DTPw-HB-Hib vaccine Administration | Baseline to 30 minutes post-vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Hung Yen, Kim Dong, Hưng Yên, Vietnam